CLINICAL TRIAL: NCT02806128
Title: The Metabolism Research of KLK Treating Acute Cerebral Ischemic Stroke: Focus on Drug Frequency-Efficacy Relationship
Acronym: MAISKFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huisheng Chen (Other)
Responsible Party: Sponsor-Investigator, Huisheng Chen, Principal Investigator, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAISKFE1.0
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-08

CONDITIONS: Cerebral Infarction
Keywords: cerebral infarction; kallikrein; KLK
MeSH Terms: conditions — Cerebral Infarction | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Injection of Human Urinary Kallidinogenase for Injection (KLK) three times a day, 14 days .
  Patients need to complete laboratory tests within a specified time.
  Interventions: Drug: Human Urinary Kallidinogenase for Injection
- Control group (Experimental): Injection of Human Urinary Kallidinogenase for Injection (KLK) Once times a day, 14 days .
  Patients need to complete laboratory tests within a specified time.
  Interventions: Drug: Human Urinary Kallidinogenase for Injection

INTERVENTIONS:
Drug: Human Urinary Kallidinogenase for Injection — Patients need to complete laboratory tests within a specified time and to complete the experimental requirements of medication time
  Other Names: KLK

SUMMARY:
Evaluate the effectiveness of the of kallikrein in the different drug frequency for acute anterior circulation cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old;
2. First time diagnosed or have history of acute anterior circulation cerebral infarction without serious sequelae (mRS = 0-2);
3. Acute anterior circulation cerebral infarction with large artery atherosclerotic etiology;
4. Ability to randomize within 48 h of time last known free of new ischemic symptoms.
5. National Institute of Health stroke scale(NIHSS) ranges from 7 to 22;
6. signed written informed consent.

Exclusion Criteria:

1. Cerebral CT shows cerebral hemorrhage disease: cerebral hemorrhage, subarachnoid hemorrhage, etc.;
2. Transient ischemic attack;
3. Serious disturbance of consciousness: Glasgow Coma ScaleGCS（GCS）≤8;
4. Combined angiotensin-converting enzyme inhibitor(ACEI) less than 5 half-time (according to its instruction), or need to be treated with ACEI;
5. Past or present suffering from hemorrhagic tendency of the disease;
6. The investigator in consideration of the other condition that the patients doesn't fit to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the decrease of National Institute of Health stroke scale(NIHSS) | 14 Days

SECONDARY OUTCOMES:
the Barthel Index | 90 Days
the Modified Rankin Scale | 90 Days
change of the National Institute of Health stroke scale | 8 Days
the composite of ischemic vascular events | 90 Days
  ischemic stroke, MI, or ischemic vascular death

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Study Chair — General Hospital of Shenyang Military Region
Locations (1):
- General hospital of shenyang military region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of clinical trials ，Through the article published and upload data 。

REFERENCES:
- [Background] Xia CF, Yin H, Borlongan CV, Chao L, Chao J. Kallikrein gene transfer protects against ischemic stroke by promoting glial cell migration and inhibiting apoptosis. Hypertension. 2004 Feb;43(2):452-9. doi: 10.1161/01.HYP.0000110905.29389.e5. Epub 2003 Dec 29. PMID 14698996
- [Background] Xia CF, Smith RS Jr, Shen B, Yang ZR, Borlongan CV, Chao L, Chao J. Postischemic brain injury is exacerbated in mice lacking the kinin B2 receptor. Hypertension. 2006 Apr;47(4):752-61. doi: 10.1161/01.HYP.0000214867.35632.0e. Epub 2006 Mar 13. PMID 16534002
- [Background] Xia CF, Yin H, Yao YY, Borlongan CV, Chao L, Chao J. Kallikrein protects against ischemic stroke by inhibiting apoptosis and inflammation and promoting angiogenesis and neurogenesis. Hum Gene Ther. 2006 Feb;17(2):206-19. doi: 10.1089/hum.2006.17.206. PMID 16454654
- [Background] Chen ZB, Huang DQ, Niu FN, Zhang X, Li EG, Xu Y. Human urinary kallidinogenase suppresses cerebral inflammation in experimental stroke and downregulates nuclear factor-kappaB. J Cereb Blood Flow Metab. 2010 Jul;30(7):1356-65. doi: 10.1038/jcbfm.2010.19. Epub 2010 Feb 24. PMID 20179726